CLINICAL TRIAL: NCT06216236
Title: Effects of Physical Fitness Using a Kinect Interventional System for Pre-frail Community-dwelling Elderly Adults
Brief Title: Effects of Physical Fitness Using a Kinect Interventional System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wan-Yun Huang (Other)
Collaborators: National Cheng Kung University (Other); Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Sponsor-Investigator, Wan-Yun Huang, Kaohsiung Veterans General Hospital, Kaohsiung Veterans General Hospital.
Organization: Kaohsiung Veterans General Hospital. (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: VGHKS20-CT4-25
Record Dates: First submitted 2023-12-29; First posted 2024-01-22 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Virtual Reality; Physical Fitness
Keywords: Physical fitness; Community dwelling elderly; Virtual reality; Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinect intervention system combined with aerobic exercise training (Experimental): Kinect intervention system combined with aerobic exercise training
  Interventions: Other: Kinect intervention system combined with aerobic exercise training; Other: aerobic dance training
- aerobic dance training (No Intervention): aerobic exercise at home.

INTERVENTIONS:
Other: Kinect intervention system combined with aerobic exercise training — A Kinect intervention system was used in the experimental group. The video displayed a skeletal simulation of the action. The participants could see their own actions and those of the teacher. After the video was completed, an accurate score for each action was displayed.
  Arms: Kinect intervention system combined with aerobic exercise training
Other: aerobic dance training — The control group used a video that did not show a skeletal simulation of the action and only saw the teachers movements.
  Arms: Kinect intervention system combined with aerobic exercise training

SUMMARY:
The Kinect intervention system combined with aerobic exercise training can improve the quality of life of older adults in the community, standardize behavior regulation in exercise and improve fitness enthusiasm.

Aerobic exercise training using the Kinect intervention system was more effective than traditional training

DETAILED DESCRIPTION:
3.3.1 Participants The subjects of this study are the elderly from the community care center in Kaohsiung City. Our goal is to recruit two groups with 30 subjects in each group, making it a total of 60 subjects. The recruitment method of this study is to upload poster advertisements in the community and the bulletin board of Kaohsiung Veterans General Hospital to recruit subjects. The purpose is to select those who meet the criteria and agree to participate in the research. Eligible subjects must sign a human experiment consent form approved by the Human Experiment Committee of Kaohsiung Veterans General Hospital.

Recruitment of subjects must meet the following standard conditions: (1) elders over the age of 65 living in the community; (2) those who use the frailty SOF scale to evaluate any of the three assessments, with the answer being "yes" for any of them (pre frailty) (given in Appendix 1); (3) able to walk independently for five minutes regardless of mobility aids; (4) drug stability in the past one month.

The exclusion criteria is as follows: (1) Those who meet the DSM-IV criteria and have psychiatric comorbidities (for example, major depression); (2) Clinically diagnosed with dementia (Dementia) or other severe cognitive impairment (mini mental state examination score less than 24 points); (3) history of stroke, traumatic brain injury or other neurological disease; (4) acute lower extremity or lower back pain, peripheral neuropathy, rheumatic- and orthopedic-related diseases; (5) unstable diseases and symptoms in the past six months, including cardiovascular disease and high blood pressure and/or diabetes; (6) those who cannot follow the exercise program or participate in other exercise programs at the same time.

All subjects who meet the inclusion conditions first fill in the general information assessment that includes basic personal characteristics, disease history, and related exercise habits. This is used to collect demographic data (depicted in Appendix 2) and fill in the Chinese version of the quality-of-life questionnaire, exercise behavior Conditioning Questionnaire, Pap Scale, Instrumental Activities of Daily Living Functioning Scale, and Mini-Mental State Test. The subject is said to have completed part of the test if they are unable to continue the remaining items due to physical and/or other factors. At this time, the subject will make an appointment to do the remaining items next time. All quizzes are expected to take approximately 40 minutes.

This study was a double-blind random assignment experiment, and the subjects and evaluators were unaware of the subjecs group. The subjects were randomly assigned to the intervention group (aerobic dance or aerobic exercise training in virtual reality), and they were asked to follow the virtual reality program to perform the requisite training. They could see whether their actions and those of other companions are correct.

The screen displays the percentage of correct movements. The time of each movement is five minutes with a 2-minute break in between for a total of 30 minutes, three times a week, for eight weeks, i.e., a total of 24 rounds. The heartbeat was monitored throughout. The control group did aerobic dance and exercise training without virtual reality. Exercise-related health education was also given, and changes in the physical functionality of the elderly living in the community were observed.

3.3.2 Intervention Aerobic dance: According to the demonstration video of the aerobic teacher, the initial training content combines basic movements with different purposes. The content is divided into 3METs, 4METs, 5METs, muscle strength training, and relaxation and stretching activity videos according to exercise intensity. Warm-up training must be done first followed by simple exercise intensity. After the task is over, a 5-minute rest is taken before entering higher-intensity task training, muscle strength training, and, finally, relaxation activities, for a total of 30 minutes.

Integrated movement training: For aerobic movement, basic activity introduction and basic movement explanation, as well as execution movement, will be analyzed by the software to find the exact ratio of movement, pulse rate, SpO2, and calories, in order to understand the basic movement training.

Circulation training: Cardiopulmonary function training uses different individuals' exercise ability and cyclic tasks as the training design. The VR training content can record the individual's usage records and exercise intensity, and perform cyclic training for individual cases, adding repetitive exercises and stimulation.

All interventions will be delivered by trained therapists, three times a week for eight weeks, with each session lasting approximately 30 minutes. Before the intervention, all subjects were screened using the Physical Activity Readiness Questionnaire (PAR-Q), and static blood pressure was checked. Those whose blood pressure was higher than 160/90 mm Hg were advised to stop the experiment. After the intervention, the subjects' breathing, heartbeat, and blood pressure were recorded to understand their physiological condition and gauge the action to be taken next. This could also involve performing primary and secondary assessment items such as physical fitness, Berg balance scale, standing time on one foot, activities of daily living,and quality of life before, immediately after, and one month after the intervention to verify the use of virtual reality aerobic dance effects of an aerobic exercise training intervention in the changes they cause in physical functionality of community-dwelling older adults.

ELIGIBILITY:
Inclusion Criteria:

* (1) individuals >60 years old who live in the community; (2) use of the SOF scale for frailty to evaluate the three assessments, any one of which satisfy the "pre-frailty" criteria; (3) able to walk independently for 5 minutes, regardless if they need a walking aid; and (4) medication usage has been stable in the past month.

Exclusion Criteria:

* (1) those with psychiatric diseases or comorbidities based on the DSM-IV criteria and had psychiatric comorbidities (e.g., major depressive disorder); (2) clinically diagnoses of dementia (dementia) or other severe cognitive impairments (Mini-Mental State Examination score <24 points); and (3) other neurological, orthopedic, and unstable diseases.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2024-02-03 (Actual); Primary Completion 2025-12-03 (Actual); Study Completion 2025-12-03 (Actual)

PRIMARY OUTCOMES:
The body mass index (BMI) | 30 min/session 3 sessions/week for 8 weeks.
  Body mass index : The formula for calculating BMI is weight (kilograms, kg) divided by height squared (meters, m2)
waist-to-hip ratio (WHR) | 30 min/session 3 sessions/week for 8 weeks.
  2 Waist-to-hip ratio (WHR) Waist circumference is an important indicator to measure abdominal obesity. Waist-to-hip ratio is one of the important indicators of obesity in the elderly, and is also a predictor of simple cardiovascular diseases. Waist measurement is taken by standing with feet shoulder-width apart using a tape measure to measure the horizontal circumference parallel to the navel;
chair stand test | 30 min/session 3 sessions/week for 8 weeks.
grip strength measurement | 30 min/session 3 sessions/week for 8 weeks.
6-minute walk (6MWT) tests | 30 min/session 3 sessions/week for 8 weeks.

SECONDARY OUTCOMES:
The Quality of Life Questionnaire by World Health Organization . | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shin-Tsu mr Chang, PhD, Study Chair — Kaohsiung Veterans General Hospital.
Locations (2):
- Taiwan (2):
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - National Cheng Kung University, Tainan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang WY, Liou IH, Chang ST, Lee CH, Du YC, Cherng RJ. Effects of physical fitness using a Kinect system for pre-frail community-dwelling older adults. Front Public Health. 2025 Jun 11;13:1498606. doi: 10.3389/fpubh.2025.1498606. eCollection 2025. PMID 40567995